CLINICAL TRIAL: NCT03775811
Title: In Vivo Computer-aided Prediction of Polyp Histology on White Light Colonoscopy
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Ana García-Rodríguez, Principal Investigator, Hospital Clinic of Barcelona
Other Study IDs: HISINVIA; PI17/00894 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2018-12-11; First posted 2018-12-14 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Colonoscopy; Histology; Computer-aided Diagnosis; Artificial Intelligence; Colorectal Polyp; Adenoma Colon Polyp; Hyperplastic Polyp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AUTOMATED POLYP CLASSIFICATION — COLONIC POLYP HISTOLOGY PREDICTION IN WHITE LIGHT IMAGES COMBINING ARTIFICIAL INTELLIGENCE AND CLINICAL INFORMATION

SUMMARY:
Our group, prior to the present study, developed a handcrafted predictive model based on the extraction of surface patterns (textons) with a diagnostic accuracy of over 90%24. This method was validated in a small dataset containing only high-quality images.

Artificial intelligence is expected to improve the accuracy of colorectal polyp optical diagnosis. We propose a hybrid approach combining a Deep learning (DL) system with polyp features indicated by clinicians (HybridAI). A pilot in vivo experiment will carried out.

DETAILED DESCRIPTION:
Optical diagnosis aims to predict the histology of a polyp based on its endoscopic features. This practice could avoid histopathological analysis and reduce the derived costs. Under this premise, the American Society of Gastrointestinal Endoscopy (ASGE), in its Preservation and Incorporation of Valuable endoscopic Innovations (PIVI) statement, established a diagnostic threshold for real-time endoscopic assessment of diminutive polyps. The rationale for its implementation is that the prevalence of advanced histology in polyps < 5mm is very low (0.5%).

Several studies have demonstrated that optical diagnosis of small polyps is safe and feasible in clinical practice and comparable to the current gold standard, histopathology. However, the accuracy of optical diagnosis has been shown to be insufficient in community-based practices or in non-expert hands and the diagnosis is even more difficult in diminutive polyps < 3 mm in which the discrepancy between the endoscopic and pathological diagnosis is about 15%.

Artificial Intelligence (AI) has emerged as a help tool for polyp characterization.

Aiming to improve optical diagnosis using AI methods, we propose a hybrid approach that combines DL with characteristics of polyps manually indicated by endoscopists (HybridAI).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Approval of participation in the study. Signature of informed consent
* Patients with at least one polyp of any size/morphology diagnosed in a routine or screening colonoscopy
* Endoscopies performed with high definition endoscopes

Exclusion Criteria:

* Age <18 years
* Refusal to participate in the study
* Polyps partially resected in a previous endoscopy
* Patients with inflammatory disease
* Impossibility to wash remains of stool or mucus on the surface of the polyp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with polyps of any size/morphology, detected in a routine or screening colonoscopy, that are resected endoscopically and recovered for histological analysis will be included.
  The images obtained will be used to expand the database.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of the computer-aided system for predicting polyps histology in real clinical practice | One year
  The results of the computer-aided system prediction will be compared with the final pathology report, which is the gold standard

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Montes C, Sanchez FJ, Bernal J, Cordova H, Lopez-Ceron M, Cuatrecasas M, Rodriguez de Miguel C, Garcia-Rodriguez A, Garces-Duran R, Pellise M, Llach J, Fernandez-Esparrach G. Computer-aided prediction of polyp histology on white light colonoscopy using surface pattern analysis. Endoscopy. 2019 Mar;51(3):261-265. doi: 10.1055/a-0732-5250. Epub 2018 Oct 25. PMID 30360010
- [Background] Bernal J, Histace A, Masana M, Angermann Q, Sanchez-Montes C, Rodriguez de Miguel C, Hammami M, Garcia-Rodriguez A, Cordova H, Romain O, Fernandez-Esparrach G, Dray X, Sanchez FJ. GTCreator: a flexible annotation tool for image-based datasets. Int J Comput Assist Radiol Surg. 2019 Feb;14(2):191-201. doi: 10.1007/s11548-018-1864-x. Epub 2018 Sep 25. PMID 30255462
- [Background] Byrne MF, Chapados N, Soudan F, Oertel C, Linares Perez M, Kelly R, Iqbal N, Chandelier F, Rex DK. Real-time differentiation of adenomatous and hyperplastic diminutive colorectal polyps during analysis of unaltered videos of standard colonoscopy using a deep learning model. Gut. 2019 Jan;68(1):94-100. doi: 10.1136/gutjnl-2017-314547. Epub 2017 Oct 24. PMID 29066576